CLINICAL TRIAL: NCT02672709
Title: Pharmacokinetics and Pharmacodynamics of Apixaban in End-stage Renal Disease Patients on Hemodialysis
Brief Title: Apixaban in Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Mark L. Lipman, Associate Professor of Medicine, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: #15-128
Record Dates: First submitted 2016-01-12; First posted 2016-02-03 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: End-stage Renal Disease
Keywords: Factor Xa Inhibitors; Renal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anticoagulation (Experimental): Apixaban will be prescribed at the dose of 2.5 mg twice per day for nine days.
  Interventions: Drug: apixaban

INTERVENTIONS:
Drug: apixaban

SUMMARY:
This study aims to determine the effects of end-stage renal disease on the pharmacokinetics, pharmacodynamics, safety, and tolerability of apixaban. This is a single-center open-label pharmacological study. Apixaban will be prescribed at the dose of 2.5 mg twice per day for nine days. The concentration of the drug will be measured with repetitive blood tests the first and the eighth day of administration (non-dialysis days). The same blood tests will be repeated before, during, and after dialysis on dialysis days. If the study shows inadequate or suboptimal efficacy with the 2.5 mg dose, it will be repeated with the 5 mg twice-daily dose.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* end-stage renal disease on stable hemodialysis treatment (3 weekly sessions of 4 hours) for at least 6 months
* no residual kidney function
* non-valvular atrial fibrillation

Exclusion Criteria:

* age ≥80 years
* Body mass index (BMI)<21 or BMI>40
* active bleeding
* high bleeding risk (HAS BLED score >3)
* active malignancy
* psychiatric disorders
* decompensated thyroid disorders
* decompensated heart failure
* acute myocardial infarction-cerebrovascular accident-head trauma in the last 3 months
* previous history of venous thromboembolic disease in the last 6 months
* previous history of coagulopathy already treated by vitamin K antagonists (VKAs) or novel oral anticoagulants
* uncorrected rhythm or conduction disturbances
* dual antiplatelet therapy
* known liver disease or elevated transaminases > 2x upper limit of normal
* Hemoglobin < 90 g/l
* platelets < 100,000 /ml
* known hypersensitivity to apixaban
* treatment with a potent inhibitor or inducer of the cytochrome P450 3A4 and/or P-glycoprotein
* absence of effective contraception where applicable
* drug or alcohol abuse

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Apixaban concentration | Day 8
  Examine whether apixaban accumulates after an 8-day administration

SECONDARY OUTCOMES:
Apixaban concentration before, during, and after hemodialysis | Before dialysis, then every hour until the end of dialysis on day 2 and day 9
  Apixaban levels to be measured before dialysis, then every hour until the end of dialysis on day 2 and day 9
Number of participants with treatment related adverse effects | Day 1 to 9
  Short-term treatment related adverse effects: bleeding events, allergic reactions, any other symptom reported by the patient that could be attributed to the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Canada

REFERENCES:
- [Background] Verma A, Cairns JA, Mitchell LB, Macle L, Stiell IG, Gladstone D, McMurtry MS, Connolly S, Cox JL, Dorian P, Ivers N, Leblanc K, Nattel S, Healey JS; CCS Atrial Fibrillation Guidelines Committee. 2014 focused update of the Canadian Cardiovascular Society Guidelines for the management of atrial fibrillation. Can J Cardiol. 2014 Oct;30(10):1114-30. doi: 10.1016/j.cjca.2014.08.001. Epub 2014 Aug 13. PMID 25262857
- [Background] Granger CB, Chertow GM. A pint of sweat will save a gallon of blood: a call for randomized trials of anticoagulation in end-stage renal disease. Circulation. 2014 Mar 18;129(11):1190-2. doi: 10.1161/CIRCULATIONAHA.113.007549. Epub 2014 Jan 22. No abstract available. PMID 24452751
- [Background] Wang X, Tirucherai G, Marbury TC, Wang J, Chang M, Zhang D, Song Y, Pursley J, Boyd RA, Frost C. Pharmacokinetics, pharmacodynamics, and safety of apixaban in subjects with end-stage renal disease on hemodialysis. J Clin Pharmacol. 2016 May;56(5):628-36. doi: 10.1002/jcph.628. Epub 2015 Dec 22. PMID 26331581